CLINICAL TRIAL: NCT01103336
Title: Preventive Effect of the PRetreatment With Intravenous Nicorandil on Contrast-Induced Nephropathy in Patients With RenaL Dysfunction UndEergoing Coronary Angiography (PRINCIPLE Study): A Investigator-initiated, Control- Randomized, Phase IV Multicenter Study
Brief Title: Preventive Effect of the PRetreatment With Intravenous Nicorandil on Contrast-Induced Nephropathy in Patients With RenaL Dysfunction UndEergoing Coronary Angiography (PRINCIPLE Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2009-0722
Record Dates: First submitted 2010-04-08; First posted 2010-04-14 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Renal Failure
Keywords: Patients with chronic renal failure undergoing coronary angiography
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicorandil in saline (Experimental)
  Interventions: Drug: pretreatment with intravenous nicorandil vs. placebo before coronary angiography
- saline (Placebo Comparator)
  Interventions: Drug: pretreatment with intravenous nicorandil vs. placebo before coronary angiography

INTERVENTIONS:
Drug: pretreatment with intravenous nicorandil vs. placebo before coronary angiography — * Nicorandil group: Pretreatment with intravenous Nicorandil (Sigmart for injection, Choongwae Pharma, Seoul) 12 mg in 0.9% saline 100 ml over 2 hours starting from 1 hour prior to coronary angiography
  * Control group: Pretreatment with intravenous 0.9% saline 100 ml over 2 hours starting from 1 hour prior to coronary angiography
  Other Names: Nicorandil group versus Control group

SUMMARY:
Renal hypoxia plays an important role in the development of contrast-induced nephropathy. The purpose of the PRINCIPLE study is to investigate the effect of pretreatment with intravenous nicorandil on the incidence of contrast-induced nephropathy in patients with renal insufficiency undergoing coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 years
* Patients undergoing elective coronary angiogram due to documented myocardial ischemia or symptoms of angina
* Estimated Cr clearance ≤60 mL/min by Cockcroft-Gault formula or serum Cr ≥1.1 mg/dL
* Signed written informed consent to participate in the study

Exclusion Criteria:

* Acute myocardial infarction requiring primary or rescue coronary intervention
* Allergic reaction to contrast dye or nicorandil
* Cardiogenic shock or significant hypotension
* Previous use of nicorandil within the preceding 7 days
* Exposure to contrast medium within the preceding 7 days
* Pregnancy or women at age of childbearing potential
* Heart failure (NYHA class III or IV; LV ejection fraction <40% by echocardiogram)
* Acute renal failure or chronic dialysis
* Mechanical ventilation
* History of kidney transplantation
* Life expectation less than 6 months
* Previous renal artery angioplasty within the last 6 months
* Use of nonsteroidal anti-inflammatory drugs, intravenous use of diuretics, dopamine, mannitol, N-acetylcysteine, ascorbic acid or sodium bicarbonate within 48 hrs before the procedure
* Severe liver disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast-induced nephropathy defined as an increase in serum creatinine ≥25% or ≥0.5 mg/dl | at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Young-Guk Ko, MD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea